CLINICAL TRIAL: NCT02659228
Title: Assessing the Potential for 'Covert Consciousness' in Unresponsive Patients
Brief Title: Assessing Covert Consciousness in Unresponsive Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Michigan (Other)
Collaborators: McGill University (Other); McMaster University (Other)
Responsible Party: Principal Investigator, George Mashour, Bert N La De Professor of Anesthesiology Research, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13-784
Record Dates: First submitted 2016-01-08; First posted 2016-01-20 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Consciousness Disorders
MeSH Terms: conditions — Consciousness Disorders | interventions — Anesthetics, Intravenous

ARMS (3):
- Control 1 (negative control) (Placebo Comparator): Individuals with a diagnosis of UWS without neural markers of consciousness
  Interventions: Device: EEG recording
- Control 2 (positive control) (Active Comparator): Individuals with a diagnosis of MCS, who are behaviourally responsive and who present neural markers of consciousness
  Interventions: Device: EEG recording
- Target Population (Experimental): Individuals with a clinical diagnosis of UWS, but who possess some neurophysiological signatures of conscious awareness
  Interventions: Device: EEG recording; Drug: Anesthetics, Intravenous

INTERVENTIONS:
Device: EEG recording — EEG recording with anesthetic (DIPRIVAN)
Drug: Anesthetics, Intravenous — The participant will receive an intravenous infusion of propofol (DIPRIVAN Injectable Emulsion USP 1%, AstraZeneca).
  Arms: Target Population

SUMMARY:
In this study, the investigators explore anesthesia as a tool for providing further insight into the level of consciousness of individuals with a clinical diagnosis of unresponsive wakefulness syndrome (UWS), but who possess some neurophysiological signatures of conscious awareness. This group, who could potentially be conscious, will herein be referred to as the target population. Our goal is to assess whether or not neurological patterns of consciousness in the target population respond to anesthesia in a similar manner to neurologically compromised individuals with known consciousness (e.g. those in minimally conscious state (MCS). In healthy controls, propofol-induced unconsciousness results in an elimination of the mismatch negativity event-related brain potential (ERP) and a diminished directed connectivity. The investigators hypothesize that at doses well below those required for surgery, anesthesia will have similar effects on these neural patterns in neurologically compromised patients with the potential for conscious awareness, but will not affect these patterns in those who lack consciousness.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the intensive care unit at Hamilton General Hospital who:

  * Clinical status consistent with UWS (no responsiveness to commands)
  * Clinical status consistent with MCS (minimal response to at least one command)
  * Presence of an endotracheal tube (ETT) or a tracheostomy tube
  * Between 18 and 50 years of age

Exclusion Criteria:

* • Elevated intracranial pressure (ICP)

  * Hepatic or renal failure
  * Hemodynamic instability
  * Active vasopressor therapy
  * Previous open-head injury
  * Previous intracranial pathology requiring neurosurgical interventions in the past 72 hours
  * Anticipated ICU stay < 24 hours
  * Documented allergy to propofol
  * Pregnancy
  * BMI > 35 kg/m2
  * Anyone who is deemed medically unsuitable for this study by the attending intensivist
  * Patients who are already in a medically-induced coma for intracranial hypertension or status epilepticus

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Asymmetry in feedback vs. feedforward network connectivity | 3 hours
  EEG networks will be monitored pre, during and post anesthesia. Directed connectivity will be calculated using phase lag index (PLI) and symbolic transfer entropy (STE) between all combinations of EEG sensors. Average values of feedback connectivity (e.g. from the frontal regions to parietal and occipital regions) will be compared to average values of feedforward connectivity (e.g. from parietal and occipital regions to frontal regions). Positive asymmetry will be correlated to the presence of conscious awareness and negative asymmetry will be correlated to the absence of conscious awareness.

SECONDARY OUTCOMES:
Presence of P300 and N400 event-related potentials | 3 hours
  EEG signals will be processed to extract the event-related EEG reactions to the auditory stimulation paradigm. Signals will be average 300 ms post-stimuli and 400 ms post-stimuli to assess the presence of the P300 and N400 event-related potentials. Presence of these event-related potentials will be correlated to the presence of conscious awareness and absence of these event-related potentials will be correlated to the absence of conscious awareness.